CLINICAL TRIAL: NCT05293249
Title: A Phase 1, Open-Label, Single Center, Dose Escalation Study of the Safety and Pharmacokinetics of mAb AZD5396 and mAb AZD8076 Delivered as dMAbs in Healthy Adults
Brief Title: dMAbs for Prevention of COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pablo Tebas (Other)
Collaborators: The Wistar Institute (Other); AstraZeneca (Industry); Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Pablo Tebas, Professor of Medicine. University of Pennsylvania, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 850355
Record Dates: First submitted 2022-03-04; First posted 2022-03-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — dMAb AZD5396; dMAb AZD8076

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (8):
- Cohort A1 - 1x 0.5 mg (Experimental): Participants (n=3) will be administered 0.5 mg of dMAb AZD5396 and 0.5 mg of dMAb AZD8076 with Hylenex® delivered intramuscularly using the side port needle followed by electroporation (EP) with OpBlock 0078 parameter on D0, for a total dose of 0.5 mg of each plasmid.
  Interventions: Combination Product: dMAb AZD5396; Combination Product: dMAb AZD8076; Combination Product: CELLECTRA™ 2000 with Side Port needle, OpBlock 0078 Electroporation device; Drug: Hylenex
- Cohort A2 - 1x 1 mg (Experimental): Participants (n=3) will be administered 1 mg of dMAb AZD5396 and 1 mg of dMAb AZD8076 with Hylenex® delivered intramuscularly using the side port needle followed by electroporation (EP) with OpBlock 0078 parameter on D0, for a total dose of 1 mg of each plasmid.
  Interventions: Combination Product: dMAb AZD5396; Combination Product: dMAb AZD8076; Combination Product: CELLECTRA™ 2000 with Side Port needle, OpBlock 0078 Electroporation device; Drug: Hylenex
- Cohort B - 2x 0.5 mg (Experimental): Participants (n=6) will be administered 0.5 mg of dMAb AZD5396 and 0.5 mg of dMAb AZD8076 with Hylenex® delivered intramuscularly using the side port needle followed by electroporation (EP) with OpBlock 0078 parameter on D0 and D3, for a total dose of 1 mg of each plasmid.
  Interventions: Combination Product: dMAb AZD5396; Combination Product: dMAb AZD8076; Combination Product: CELLECTRA™ 2000 with Side Port needle, OpBlock 0078 Electroporation device; Drug: Hylenex
- Cohort C - 2x 1 mg (Experimental): Participants (n=6) will be administered 1mg of dMAb AZD5396 and 1 mg of dMAb AZD8076 with Hylenex® delivered intramuscularly using the side port needle followed by electroporation (EP) with OpBlock 0078 parameter on D0 and D3, for a total dose of 2 mg of each plasmid.
  Interventions: Combination Product: dMAb AZD5396; Combination Product: dMAb AZD8076; Combination Product: CELLECTRA™ 2000 with Side Port needle, OpBlock 0078 Electroporation device; Drug: Hylenex
- Cohort D - 2x 0.25 mg (Experimental): Participants (n=6) will be administered 1 mg of dMAb AZD5396 and 1 mg of dMAb AZD8076 with Hylenex® delivered intramuscularly using the side port needle followed by electroporation (EP) with OpBlock 0078 parameter on D0 and D3, for a total dose of 2 mg of each plasmid.
  Interventions: Combination Product: dMAb AZD5396; Combination Product: dMAb AZD8076; Combination Product: CELLECTRA™ 2000 with Side Port needle, OpBlock 0078 Electroporation device; Drug: Hylenex
- Cohort E - 2x 2 mg (Experimental): Participants (n=5) will be administered 2 mg of dMAb AZD5396 and 2 mg of dMAb AZD8076 with Hylenex® delivered intramuscularly using the side port needle followed by electroporation (EP) with OpBlock 0078 parameter on D0 and D3, for a total dose of 4 mg of each plasmid.
  Interventions: Combination Product: dMAb AZD5396; Combination Product: dMAb AZD8076; Combination Product: CELLECTRA™ 2000 with Side Port needle, OpBlock 0078 Electroporation device; Drug: Hylenex
- Cohort F - 2x 0.5 mg (Experimental): Participants (n=5) will be administered 0.5 mg of dMAb AZD5396 and 0.5 mg of dMAb AZD8076 with Hylenex® delivered intramuscularly using the side port needle followed by electroporation (EP) with OpBlock 0070 parameter on D0 and D3, for a total dose of 1 mg of each plasmid.
  Interventions: Combination Product: dMAb AZD5396; Combination Product: dMAb AZD8076; Drug: Hylenex; Combination Product: CELLECTRA™ 2000 with Side Port needle, OpBlock 0070 Electroporation device
- Cohort G - 4x 0.5 mg (Experimental): Participants (n=5) will be administered 0.5 mg of dMAb AZD5396 and 0.5 mg of dMAb AZD8076 with Hylenex® delivered intramuscularly using the side port needle followed by electroporation (EP) with OpBlock 0078 parameter on D0, D3, D28 and D31, for a total dose of 2 mg of each plasmid.
  Interventions: Combination Product: dMAb AZD5396; Combination Product: dMAb AZD8076; Combination Product: CELLECTRA™ 2000 with Side Port needle, OpBlock 0078 Electroporation device; Drug: Hylenex

INTERVENTIONS:
Combination Product: dMAb AZD5396 — Participants will receive one injection of dMAb AZD5396 with Hylenex into the arm (deltoid)/leg (quadriceps) region followed by EP.
Combination Product: dMAb AZD8076 — Participants will receive one injection of dMAb AZD8076 with Hylenex into the arm (deltoid)/leg (quadriceps) region followed by EP.
Combination Product: CELLECTRA™ 2000 with Side Port needle, OpBlock 0078 Electroporation device — The device will be used to perform electroporation (EP) on each subject immediately after being dosed with dMAb AZD5396 and dMAb AZD8076.
  Arms: Cohort A1 - 1x 0.5 mg; Cohort A2 - 1x 1 mg; Cohort B - 2x 0.5 mg; Cohort C - 2x 1 mg; Cohort D - 2x 0.25 mg; Cohort E - 2x 2 mg; Cohort G - 4x 0.5 mg
Drug: Hylenex — Hylenex® recombinant will be used for dMAb AZD5396 and dMAb AZD8076 dose preparation at the clinical site.
Combination Product: CELLECTRA™ 2000 with Side Port needle, OpBlock 0070 Electroporation device — The device will be used to perform electroporation (EP) on each subject immediately after being dosed with dMAb AZD5396 and dMAb AZD8076.
  Arms: Cohort F - 2x 0.5 mg

SUMMARY:
This is a Phase 1, open-label, single center, dose escalation study to evaluate the safety, tolerability and pharmacokinetic profile of mAb AZD5396 and mAb AZD8076 following delivery of optimized dMAb AZD5396 and dMAb AZD8076 with Hylenex® Recombinant, administered by intramuscular injection (IM) followed immediately by electroporation (EP) using the CELLECTRA™ 2000 with Side Port needle device, in a 2-dose regimen (Days 0 and 3) or a 4-dose regimen (Days 0, 3, 28 and 31) in healthy adults.

The hypothesis is that the administration of dMAb AZD5396 and dMAb AZD8076 will be safe and associated with expression of mAb AZD5396 and mAb AZD8076 in serum.

DETAILED DESCRIPTION:
The study will apply a single ascending dose (SAD) modified 3+3 design. Participants will be enrolled sequentially beginning with Cohort A1. The first participant in cohort A1 will be dosed on Day 0. If no stopping event (DLT) is observed after 14 days of the initial dose, the remaining two participants in that cohort will be dosed. If there are 0 DLT events after 14 days of the initial dosing of the third subject, enrollment will be completed, and then cohort A2 will open. Same process will be followed for Cohorts B, C and E. Because cohorts D, F & G are a similar or lower dose and the safety profile would have been already established in previous cohorts, the 14-day waiting periods will not apply to Cohorts D, F or G.

If one dose limiting toxicity (DLT) is observed in the first three participants enrolled in any cohort, an ad hoc DSMB will review the event and make a decision if the study should continue. If the DSMB agrees that the study should continue, the remaining participants will be enrolled in the cohort and dosed, but the next cohort will not open until the 28-day period of safety is completed. However, if any additional DLT occurs (i.e., >1 DLT in 6 total participants in a given cohort), then that dose will be deemed not tolerated

The following Investigational product administration- and/or EP-related adverse events are defined as DLTs:

* Grade 3 or greater local injection site erythema, swelling, and/or induration recorded ≥ 1 hour after Investigational product administration
* Pain or tenderness at the injection site that requires overnight hospitalization despite proper use of non-narcotic analgesics.
* Grade 3 or greater systemic symptoms assessed by the Principal Investigator as related to Investigational product administration.
* Grade 3 or greater clinically significant laboratory abnormalities assessed by the Principal Investigator as related to Investigational product administration.

ELIGIBILITY:
Inclusion Criteria

1. Age 18-60 years.
2. Able to provide consent to participate and having signed an Informed Consent Form (ICF).
3. Able and willing to comply with all study procedures.
4. Body mass index (BMI) between 20 and 31, inclusive.
5. Screening laboratory must be within normal limits or have only Grade 0-1 findings.
6. Normal screening ECG or screening ECG with no clinically-significant findings.
7. Women of child-bearing potential agree to one of the following:

   1. use medically effective contraception (oral contraception, barrier methods, spermicide, etc.)
   2. have a partner who is sterile from enrollment to 6 months following the last injection
   3. have a partner who is medically unable to induce pregnancy Abstinence is acceptable per Investigator discretion and as long as it is documented that the subject will use medically effective contraception when engaging in sexual activities and notifies the study team.
8. Sexually active men who are considered sexually fertile must agree to one of the following:

   1. use a barrier method of contraception during the study and continue its use for at least 6 months following the last injection
   2. have a partner who is permanently sterile or is medically unable to become pregnant
9. No history of clinically significant immunosuppressive or autoimmune disease. Individuals with HIV infection who have been virologically suppressed for more than 1 year and with current CD4 cell count entry greater than 500 cells/ul will be allowed into the study.

Exclusion Criteria

1. Administration of an investigational compound either currently or within 6 months of first dose.
2. Administration of any vaccine within 4 weeks of first dose.
3. Administration of a SARS-CoV-2 vaccine in the last 14 days or plans to have any standard of care vaccines within 14 days form the last administration of study products.
4. Positive SARS-CoV-2 infection at screening visit.
5. Administration of any monoclonal or polyclonal antibody product within 4 weeks of the first dose.
6. Administration of any blood product within 3 months of first dose.
7. Co-morbid conditions including poorly-controlled diabetes (HbA1C > 7), poorly-controlled hypertension (BP > 140/95 repeatedly), asthma, and any cardiovascular disease.
8. Pregnancy or breast feeding or plans to become pregnant during the course of the study.
9. Positive serologic test for hepatitis B surface antigen (HBsAg); or any potentially communicable infectious disease as determined by the Principal Investigator or Medical Director.
10. Positive serologic test for hepatitis C (exception: successful treatment with confirmation of sustained virologic response);
11. Baseline evidence of kidney disease as measured by creatinine greater than 1.5 mg/dL (CKD Stage II or greater);
12. Baseline screening lab with Grade 2 or higher abnormality, except for Grade 2 creatinine.
13. Chronic liver disease or cirrhosis.
14. Immunosuppressive illness including hematologic malignancy, history of solid organ or bone marrow transplantation.
15. Current or anticipated concomitant immunosuppressive therapy (inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or prednisone at a dose less than 10 mg/day or steroid dose-equivalent are not exclusionary).
16. Current or anticipated treatment with TNF-α inhibitors such as infliximab, adalimumab, etanercept.
17. Prior major surgery or any radiation therapy within 6 months of first dose.
18. Any pre-excitation syndromes, e.g., Wolff-Parkinson-White syndrome.
19. Presence of a cardiac pacemaker or automatic implantable cardioverter defibrillator (AICD)
20. Fewer than two acceptable sites available for IM injection and EP considering the deltoid and anterolateral quadriceps muscles. The following are unacceptable sites:

    1. Tattoos, keloids or hypertrophic scars located within 2 cm of intended administration site.
    2. Implantable-Cardioverter-defibrillator (ICD) or pacemaker (to prevent a life-threatening arrhythmia) that is located ipsilateral to the deltoid injection site (unless deemed acceptable by a cardiologist).
    3. Any metal implants or implantable medical device within the electroporation site.
21. Prisoner or participants who are compulsorily detained (involuntary incarceration) for treatment of either a physical or psychiatric illness.
22. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements or assessment of immunologic endpoints.
23. Not willing to allow storage and future use of samples for SARS-CoV-2 virus related research.
24. Any illness or condition that in the opinion of the investigator may affect the safety of the participant or the evaluation of any study endpoint.
25. Participants with known bleeding diatheses or that are using blood thinners for 30 days before study enrollment including warfarin, heparin, Clopidogrel, Apixaban (Eliquis), Dabigatran (Pradaxa), Edoxaban (Savaysa), Rivaroxaban (Xarelto). The use of low dose aspirin (81 mg daily) is acceptable.
26. Participants with concomitant intramuscular medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Frequency and nature of injection site reaction | 7 days after administration of the investigational products
  Injection site reactions occurring up to 7 days after administration of the investigational product
Frequency and nature of systemic reactions | 7 days after administration of the investigational products
  Systemic reactions occurring up to 7 days after administration of the investigational product.
Frequency and nature of Serious Adverse Events | 72 Weeks after administration of the investigational products
  SAE will be classified using the CTCAE v5 throughout the study
Evaluation of the pain experienced by the participant | Immediately after EP, 5 minutes after EP and 10 minutes after EP
  Visual analogue scale (VAS). A VAS consists of a horizontal line, 10 cm in length, anchored by word descriptors at each end (no pain = 0 cm; worst pain = 10 cm). The VAS score is determined by measuring in centimeters from the left hand end of the line to the point that the patient marks. Absolute initial value and change over time will be described.
Evaluation of laboratory related adverse events | Up to 7 days after administration of the investigational product
  Laboratory AEs will be assessed and graded in accordance with the "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials", issued in September 2007.
Serum concentration of dMAb AZD5396 nm/mL. | Up to 72 Weeks after administration of the investigational products
  The number and percentage of participants in which detection of monoclonal antibody dMAb AZD5396 in serum is achieved will be summarized with a point estimate and corresponding exact 90% Clopper- Pearson confidence interval. These will be summarized per time point within each cohort. We will also estimate the time to 50% decline from peak concentration.
Serum concentration of dMAb AZD8076 nm/mL. | Up to 72 Weeks after administration of the investigational products
  The number and percentage of participants in which detection of monoclonal antibody dMAb AZD8076 in serum is achieved will be summarized with a point estimate and corresponding exact 90% Clopper- Pearson confidence interval. These will be summarized per time point within each cohort. We will also estimate the time to 50% decline from peak concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Tebas P, Patel A, Agnes JT, Parzych EM, Baer A, Caturla M, Ghosh S, Purwar M, Bedanova N, Tsang C, Morales K, Amante D, Fisher PD, Francica JR, Humeau L, Kulp DW, Pallesen J, Leon P, Esser M, Smith TRF, Weiner DB. Safety and pharmacokinetics of SARS-CoV-2 DNA-encoded monoclonal antibodies in healthy adults: a phase 1 trial. Nat Med. 2025 Dec;31(12):4150-4159. doi: 10.1038/s41591-025-03969-0. Epub 2025 Oct 21. PMID 41120767

DOCUMENTS (1):
  • Informed Consent Form (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT05293249/ICF_000.pdf